CLINICAL TRIAL: NCT02672280
Title: Safety and Exploratory Efficacy Study of Collagen Membrane With Mesenchymal Stem Cells in the Treatment of Skin Defects
Acronym: SEESCMMSCTSD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-3
Record Dates: First submitted 2016-01-31; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Wounds; Diabetic Foot Ulcers; Burns
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot; Burns

ARMS (2):
- Medical Collagen Membrane with MSC (Experimental): Applications of medical collagen membrane with umbilical cord derived mesenchymal stem cells (MSC).
  Interventions: Device: Medical Collagen Membrane with MSC
- Medical Collagen Membrane (Active Comparator): Application of medical collagen membrane only.
  Interventions: Device: Medical Collagen Membrane

INTERVENTIONS:
Device: Medical Collagen Membrane with MSC
  Arms: Medical Collagen Membrane with MSC
Device: Medical Collagen Membrane
  Arms: Medical Collagen Membrane

SUMMARY:
The purpose of the present study is to evaluate the safety and exploratory efficacy of the medical collagen membrane with umbilical cord derived mesenchymal stem cells in the treatment of patients with skin defects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70, borh gender.
* Patient able and willing to sign informed consent and comply with study procedures.
* Women of childbearing potential must use birth control pills, barriers or abstinence and have a negative pregnancy test.
* Deep partial or full thickness skin defect of at least 9 cm2 requiring surgical wound coverage due to: burn injury, diabetic foot ulcer or wounds caused by mechanical damage or iatrogenic injury.

Exclusion Criteria:

* Patient refusal.
* Patient has a documented history of allergy or sensitivity to any of the animal products used in preparation of skin substitute. These products include bovine blood, bovine collagen, and bovine collagenase.
* Patient has a documented history of allergy or sensitivity to any of the antimicrobials or reagents used in preparation and application of skin substitute including the irrigation solution used before and after grafting.
* Patient has a current diagnosis of an invasive burn wound infection in unexcised burn wound.
* Patient has tunnels or sinus tracts that cannot be completely debrided.
* Serious primary diseases of the liver, kidney and hematopoietic system, Abnormal liver function(glutamic-pyruvic transaminase(ALT), glutamicoxalacetic transaminase (AST) is 2 times higher than the normal value), creatinine(Cr) is higher than the upper limit of the normal value.
* Other clinical trial participants within 3 months.
* A random blood sugar reading >/=450 mg/dL.
* Investigators judge other conditions not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events that are related to study treatment and associated with the grafting site | Up to Month 36 after the last grafting day
Percentage of wound closure as determined | Up to Month 3 after the last grafting day

SECONDARY OUTCOMES:
Scar outcome assessment | Up to Month 36 after the last grafting day
Incidence of contracture release or revision surgeries | Up to Month 36 after the last grafting day
Incidence of increased temperature sensitivity | Up to Month 36 after the last grafting day
Incidence of paresthesias, pain, dulling of sensation assessed | Up to Month 36 after the last grafting day
Incidence and severity of infections at grafting sites | Up to Month 6 after the last grafting day
Incidence of all adverse events | Up to Month 36 after the last grafting day
Percentage area of re-grafting as determined | Up to Month 6 after the last grafting day

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He L, Nan X, Wang Y, Guan L, Bai C, Shi S, Yuan H, Chen L, Liu D, Pei X. Full-thickness tissue engineered skin constructed with autogenic bone marrow mesenchymal stem cells. Sci China C Life Sci. 2007 Aug;50(4):429-37. doi: 10.1007/s11427-007-0069-2. PMID 17653662
- See also: Related Info — http://link.springer.com/article/10.1007%2Fs11427-007-0069-2